CLINICAL TRIAL: NCT06088953
Title: DEAFNESS SCREENING IN A MEMORY CENTER IN SUBJECTS WITH COGNITIVE DISORDERS
Brief Title: EARLY DETECTION OF DEAFNESS IN A MEMORY CENTER
Acronym: CogAudio
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2022_0392
Record Dates: First submitted 2023-08-21; First posted 2023-10-18 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Cognitive Disorder; Deafness
Keywords: Cognitive Disorder; Deafness
MeSH Terms: conditions — Cognitive Dysfunction; Deafness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- perception disorder in noise in patients weakened by cognitive disorders. (Experimental): The CogAudio project aims to detect early and in an ambulatory mode in a memory centre a speech perception disorder in noise thanks to the VRB test in patients weakened by cognitive disorders.
  Interventions: Diagnostic Test: VRB test

INTERVENTIONS:
Diagnostic Test: VRB test — V1 (inclusion) : VRB test for detecting speech comprehension disorders in noise.
  V2 (3 months) : all patients ( independent of the result of the VRB test) will be invited to attend a hearing test within 3 months in order to confirm the diagnosis of deafness by means of a tone audiometry and an ENT medical consultation.

SUMMARY:
Age-related hearing loss (ARHL), like neurodegenerative diseases, appears insidiously with age. As major public health issues, they are nonetheless under-diagnosed because the presence of one can hinder the objectification of the other.

The CogAudio project aims to detect early and in an ambulatory mode in a memory centre a speech perception disorder in noise thanks to the VRB test in patients weakened by cognitive disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patient with mild to moderate cognitive impairment, with an MMSE score ≥15/30
* Patient mastering the French language
* Patient who has given written consent to participate in the trial
* Socially insured patient
* Patient willing to comply with all study procedures and duration
* Patient accompanied by a study partner

Exclusion Criteria:

* Medical history of diagnosed deafness, fitted or not
* History of progressive otological pathology or presence of tympanic obstruction (>1/3 of the surface of the eardrum)
* History of unstabilized psychiatric pathology
* Major visual impairment (Age-Related Macular Degeneration AMD...)
* Established diagnosis of major language disorders (Primary Progressive Aphasia APP...)
* Major under legal protection measure

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2026-08-27 (Estimated); Study Completion 2027-08-27 (Estimated)

PRIMARY OUTCOMES:
Ability of the VRB test to detect deafness in patients over 50 with mild to moderate cognitive impairment. | 3 months
  Area under the ROC (receiver operating characteristic) curve of the VRB test for hearing loss screening.

SECONDARY OUTCOMES:
To assess the diagnostic values of the VRB threshold associated with a disorder of speech comprehension in noise defined in the general population to screen for deafness in patients over 50 years of age with mild to moderate cognitive impairment. | 3 months or 12 months
  Sensitivity, specificity, negative and positive predictive values of the pathological threshold defined in the general population (>3 BSR ) for hearing loss screening (as defined in the primary endpoint)
correlation between the hearing loss and the auditory discomfort (complaint) expressed by the patient and that observed by the caregiver | 3 months or 12 months
  Hearing loss is defined by the VRB test score. The auditory complaint expressed by the patient is defined by the score on the HHIE-S questionnaire completed by the patient himself; the auditory complaint noted by the entourage is defined by the score on the adapted HHIE-S questionnaire completed by the caregiver present at the consultation at M0.
Frequency of patients with hearing aids at 12 months. | 3 months or 12 months
  Frequency of patients with hearing aids at 12 months from inclusion
Evolution of the cognitive and functional profile at 12 months between patients with deafness and patients without deafness. | 3 months or 12 months
  Variation in scores between M0 and M12 on HAD neuropsychological and speech therapy test.
To assess the correlation between an objective cortical marker of selective attention (long latency evoked potentials: P300 wave amplitude; patients' ability to discriminate sounds in silence), and subjects' performance in tone audiometry in silence | 3 months or 12 months
  Amplitude and latency of the P300 wave; Tone audiometry score in silence.
Evolution of the cognitive and functional profile at 12 months between patients with deafness and patients without deafness. | 3 months or 12 months
  Variation in scores between M0 and M12 on WHOQOL-BREF neuropsychological test
Evolution of the cognitive and functional profile at 12 months between patients with deafness and patients without deafness. | 3 months or 12 months
  Variation in scores between M0 and M12 on QFS functional scale
Evolution of the cognitive and functional profile at 12 months between patients with deafness and patients without deafness. | 3 months or 12 months
  Variation in scores between M0 and M12 on LARS neuropsychological test.
Evolution of the cognitive and functional profile at 12 months between patients with deafness and patients without deafness. | 3 months or 12 months
  Variation in scores between M0 and M12 on EQ-5D-3L neuropsychological test.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Roger Salengro, Lille, France

IPD SHARING:
Plan to Share IPD: No